CLINICAL TRIAL: NCT02709148
Title: State-dependent Pathophysiological Oscillations in Parkinson's Disease and Treatment With DBS
Brief Title: State-dependent Pathophysiological Oscillations in Parkinson's Disease and Treatment With Deep Brain Stimulation (DBS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NEURO-2016-24512
Record Dates: First submitted 2016-03-01; First posted 2016-03-15 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- chronic brain recording (Experimental): This is a one-arm, single-center study of the neurophysiology of human movement disorders with two goals: 1) Assess the feasibility of chronic brain recording using a novel fully implantable pulse generator (Medtronic Activa PC+S), which has the capability of sensing and storing local field potentials (LFPs) recorded from implanted electrodes, in addition to providing therapeutic deep brain stimulation (DBS). 2) Study acute and chronic effects of therapeutic DBS on cortical LFPs. 3) Study feasibility of the use of brain signals as feedback either directly to the patient or for DBS stimulation adjustments.
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — DBS

SUMMARY:
The purpose of this study is to use an investigational device to record brain activity for 12-24 months following surgical implantation of deep brain stimulation (DBS) systems. The goal of the study is better understanding of brain activity in Parkinson's disease and how they relate to DBS and pharmacological management, not to bring new devices to market.

DETAILED DESCRIPTION:
Experimental: chronic brain recording This is a one-arm, single-center study of the neurophysiology of human movement disorders with two goals: 1) Assess the feasibility of chronic brain recording using a novel fully implantable pulse generator (Medtronic Activa PC+S), which has the capability of sensing and storing local field potentials (LFPs) recorded from implanted electrodes, in addition to providing therapeutic deep brain stimulation (DBS). 2) Study acute and chronic effects of therapeutic DBS on cortical LFPs. 3) Study feasibility of the use of brain signals as feedback either directly to the patient or for DBS stimulation adjustments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's Disease (PD).
2. Age 45-75 years
3. UPDRS III motor score (off PD medications) ≥ 25
4. Demonstrated good response (≥ 30%) to Sinemet or dopamine agonist medications as assessed by total UPDRS III score (off and on meds)
5. Approved for unilateral subthalamic nucleus (STN)- or globus pallidus internus (GPi)-DBS surgery to treat their clinical motor signs and plan to undergo the standard of care procedure within the next four months
6. Cleared to be scanned in a 7 tesla magnet
7. Written documentation of willingness to participate in the study per protocol as evidenced by the informed consent process

Exclusion Criteria:

1. Clinically significant medical disease that would increase the risk of developing pre- or post-operative complications (e.g., significant cardiac or pulmonary disease)
2. Evidence of secondary or atypical parkinsonism
3. Dementia as evidenced by impairment in two neuropsychological domains and impaired or borderline neuropsychological function in one additional domain.
4. Unable to undergo magnetic resonance imaging (e.g., due to incompatible implanted pacemaker)
5. Previous pallidotomy or DBS surgery
6. Women who are currently pregnant or are breast feeding
7. MRI showing cortical atrophy out of proportion to age and/or MRI showing focal brain lesions that could indicate a non-idiopathic movement disorder
8. Any prior intracranial surgery
9. Subjects with depression defined according to Diagnostic and Statistical Manual V criteria and a scored on a validated depression assessment scale
10. History of seizures
11. Immunocompromised
12. Requires diathermy, electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) to treat a chronic condition
13. Has an implanted electronic device such as a neurostimulator, cardiac pacemaker or medication pump.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Cortical and sub-cortical brain signals using Activa PC+S | 12 months
  Establish whether it is possible to record a reliable cortical and subcortical brain signal using Activa PC+S.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Vitek, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided